CLINICAL TRIAL: NCT03975491
Title: The Exercise And Colorectal Cancer Treatment (EXACT) Trial
Brief Title: The Exercise And Colorectal Cancer Treatment Trial
Acronym: EXACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Justin Brown, Adjunct Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2019-009; R00CA218603 (NIH)
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Moderate-intensity aerobic exercise
  Interventions: Behavioral: Moderate-Intensity Aerobic Exercise
- Control (Sham Comparator): Wait-list control
  Interventions: Behavioral: Wait-List Control

INTERVENTIONS:
Behavioral: Moderate-Intensity Aerobic Exercise — The exercise intervention will consist of moderate-intensity (50-70% age-predicted maximum heart rate) treadmill walking. All exercise sessions will begin with a five-minute warm up of slow walking, 30-60 minutes of moderate-intensity walking, and a five-minute cool down of slow walking.
  Arms: Aerobic Exercise
Behavioral: Wait-List Control — Participants randomized into the wait-list control group are asked to maintain their pre-study levels of physical activity and follow the recommendations provided by their physician.
  Arms: Control

SUMMARY:
This study will examine the biologic processes through which exercise may prevent disease recurrence in patients who have completed treatment for colorectal cancer.

DETAILED DESCRIPTION:
This randomized trial will examine the biological effects of 12-weeks of moderate-intensity aerobic exercise versus wait-list control in 60 subjects who have completed standard medical therapy for colorectal cancer. The primary objective is to determine if aerobic exercise can reduce systemic inflammation, quantified using plasma concentrations of high-sensitivity C-reactive protein and interleukin-6. The secondary objectives are to determine if exercise can reduce: 1) insulin resistance quantified using an oral glucose tolerance test, and; 2) circulating tumor cells quantified using a microfluidic antibody-mediated capture platform. The exploratory objective is to determine if exercise can improve mitochondrial respiration rates and fatty acid oxidation in peripheral blood mononuclear cells and tumor fraction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically-confirmed stage I-III colorectal cancer
* Completed surgical resection
* Completed chemotherapy (if applicable)
* Completed radiotherapy (if applicable)
* Provide written approval by physician or other qualified healthcare provider
* No planned major surgery during the study period (including colostomy reversal; chemotherapy infusion port removal is permitted)
* Readiness to exercise [as determined by a modified version the Physical Activity Readiness Questionnaire (PAR-Q)
* Allow the collection and storage of specimens and data for future use
* Willing to be randomized

Exclusion Criteria:

* Evidence of metastatic colon cancer
* Concurrently actively treated other cancer (except non-melanoma skin cancer or in situ cancers)
* Currently enrolled in another clinical trial of weight loss, physical activity, or dietary intervention
* Current body mass greater than or equal to 181 kg
* Unable to provide a baseline fasting blood sample
* Unable or unwilling to give informed consent
* Unable or unwilling to be randomized
* Or any other condition that may impede testing of the study hypothesis or make it unsafe to engage in the exercise program (as determined by the investigative team)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2026-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Justin C Brown, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reporting and publication of the primary, secondary, and exploratory study outcomes de-identified individual participant data will be released to investigators.
Supporting Information: Study Protocol, SAP
Time Frame: After reporting and publication of the primary, secondary, and exploratory study outcomes is complete.
Access Criteria: Data will be shared according to the principles outlined by Tudur Smith et al in BMC Medicine 2015.

REFERENCES:
- [Background] Compton SLE, Yang S, Maniscalco LS, Muhsen RA, Shrestha P, Wu X, Woodard KT, Zunica ERM, Cho E, Wall RL, Brown J, Jayaraman A, Kirby BJ, Gilmore LA, Greenway FL, Spielmann G, Brown JC. A randomized trial of aerobic exercise in colorectal cancer: Rationale, design, recruitment, and exercise adherence results. Contemp Clin Trials. 2024 Nov;146:107702. doi: 10.1016/j.cct.2024.107702. Epub 2024 Oct 1. PMID 39362405
- [Background] Cho E, Chodzko M, Compton SLE, Yang S, Heymsfield S, Spielmann G, Brown JC. Effects of aerobic exercise on body composition and exerkines in colorectal cancer survivors. Front Sports Act Living. 2025 Jun 26;7:1579221. doi: 10.3389/fspor.2025.1579221. eCollection 2025. PMID 40642656
- [Result] Brown JC, Compton SLE, Kang A, Jayaraman A, Gilmore LA, Kirby BJ, Greenway FL, Yang S, Spielmann G. Effects of exercise on inflammation, circulating tumor cells, and circulating tumor DNA in colorectal cancer. J Sport Health Sci. 2025 Dec;14:101036. doi: 10.1016/j.jshs.2025.101036. Epub 2025 Mar 17. PMID 40107449

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: Aerobic Exercise
- Control: Waitlist Control
Period: Overall Study
Arm/Group | Exercise | Control
Started | 31 | 29
Completed | 31 | 28
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Control | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.9) | 58.6 (10.6) | 60.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 39
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
High Sensitivity C-Reactive Protein [Geometric Mean (Standard Deviation); unit: mg/L] | 2.6 (2.1) | 2.4 (2.2) | 2.5 (2.1)
Interleukin-6 [Geometric Mean (Standard Deviation); unit: pg/mL] | 6.2 (4.2) | 3.8 (3.9) | 4.8 (4.1)
Soluble Tumor Necrosis Factor-Alpha Receptor Two [Geometric Mean (Standard Deviation); unit: pg/mL] | 6307.7 (1.4) | 5598.5 (1.4) | 5954.4 (1.5)
Circulating Tumor Cells [Mean (Standard Deviation); unit: cells/mL] | 1.6 (1.9) | 1.5 (2.2) | 1.5 (2.0)
Tumor Fraction [Mean (Standard Deviation); unit: % cells of tumor origin (of all cfDNA)] | 0.009 (0.003) | 0.012 (0.009) | 0.010 (0.007)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in High-sensitivity C-reactive Protein
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Exercise | Control
Number analyzed (Participants) | 31 | 28
% change | 12.8 [-13.1 to 46.3] | -6.7 [-28.9 to 22.4]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Net) = 20.9, 95% CI 2-sided [-17.1 to 76.2] — From a model that included the baseline value of the dependent variable and sex (randomization stratification factor) as covariates

2. Primary Outcome: The Percentage Change in Interleukin-6
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Exercise | Control
Number analyzed (Participants) | 31 | 28
% change | -15.0 [-25.4 to -3.2] | -5.4 [-17.0 to 7.9]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Net) = 11.4, 95% CI 2-sided [-7.5 to 34.0] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: The Percentage Change in Soluble Tumor Necrosis Factor-alpha Receptor Two
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Exercise | Control
Number analyzed (Participants) | 31 | 28
% change | -2.1 [-9.3 to 5.7] | 1.6 [-6.2 to 10.0]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.52, Mixed Models Analysis; Mean Difference (Net) = -3.6, 95% CI 2-sided [-13.7 to 7.7] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: The Change in Circulating Tumor Cells Per mL Whole Blood
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: cells/mL
Arm/Group | Aerobic Exercise | Control
Number analyzed (Participants) | 31 | 28
cells/mL | -0.02 [-0.56 to 0.52] | -0.61 [-1.36 to 0.14]
Statistical Analysis 1: Comparison: Aerobic Exercise vs Control; Test type: Superiority; p = 0.21, Mixed Models Analysis; Mean Difference (Net) = 0.59, 95% CI 2-sided [-0.33 to 1.51] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Insulin Resistance
Description: Oral Glucose Tolerance Test (2 hour AUC)
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

6. Other Pre Specified Outcome: The Percentage Change in Circulating Tumor DNA (Relative to All Cell-free DNA)
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: % change
Arm/Group | Exercise | Control
Number analyzed (Participants) | 31 | 28
% change | 0.0011 [-0.0009 to 0.0031] | 0.0006 [-0.0015 to 0.0027]
Statistical Analysis 1: Comparison: Exercise vs Control; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Net) = 0.0005, 95% CI 2-sided [-0.0024 to 0.0034] — [estimate comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Mitochondrial Respiration Rate
Description: Respiration rate in peripheral blood mononuclear cells (pmol O2/sec/million cells)
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

8. Other Pre Specified Outcome: Fatty Acid Oxidation
Description: Oxidation rate in peripheral blood mononuclear cells (mmol/mg/min)
Time Frame: Baseline, 12 weeks
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

LIMITATIONS AND CAVEATS:
Results of other endpoints not submitted on July 25, 2025, will be reported at a later date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03975491/Prot_SAP_000.pdf